CLINICAL TRIAL: NCT03641105
Title: Investigation of the Contents and Prognostic Values of Glucose Metabolism Molecules in Patients With Lung Adenocarcinoma
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ZST-GLUMETA
Record Dates: First submitted 2018-08-18; First posted 2018-08-21 (Actual); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Lung Cancer; Glycolysis; Diagnosis; Survival
MeSH Terms: conditions — Lung Neoplasms; Disease | interventions — Diagnostic Tests, Routine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- lung adenocarcinoma: patients with lung adenocarcinoma
  Interventions: Diagnostic Test: Diagnostic test

INTERVENTIONS:
Diagnostic Test: Diagnostic test — detect the contents of glucose metabolism molecules using mass spectrum

SUMMARY:
Detect the contents of glucose metabolism molecules in the tumor and adjacent normal samples of about 100 patients with lung adenocarcinoma using mass spectroscopy. Analyze the correlation between the contents and the clinicopathological characteristics and survival.

ELIGIBILITY:
Inclusion Criteria:

* Primary lung adenocarcinoma

Exclusion Criteria:

* Other tumor histories, received radiotherapy or chemotherapy before surgery, tumor or adjacent normal tissues can't be obtained, patient rejected.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with primary lung adenocarcinoma
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2014-01-01 (Actual); Primary Completion 2019-03-01 (Estimated); Study Completion 2019-03-01 (Estimated)

PRIMARY OUTCOMES:
disease-free survival | 1 month
  disease-free survival

SECONDARY OUTCOMES:
overall survival | 1 month
  overall survival